CLINICAL TRIAL: NCT06545695
Title: Epidermal Growth Factor Receptor Inhibition for Keratinopathies
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP08062024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: Epidermolytic Ichthyosis; Palmoplantar Keratoderma; Pachyonychia Congenita
MeSH Terms: conditions — Hyperkeratosis, Epidermolytic; Keratoderma, Palmoplantar; Pachyonychia Congenita | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Erlotinib Treatment Arm (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Part B will be the dose escalation component, in which the subject will initiate 50 mg erlotinib,8 weeks later escalate to 75 mg, and then 8 weeks later to 100 mg erlotinib pending tolerance after each 8-week period.

SUMMARY:
Epidermal growth factor receptor (EGFR) signaling plays a key role in regulating epidermal cell proliferation, survival, and differentiation. Keratins form a scaffold with epidermal desmosomes that involves ErbB/ EGFR signaling and keratin deficiency makes keratinocytes more sensitive to EGFR activation. Erlotinib, an EGFR inhibitor, was approved 20 years ago for cancer treatment and is generally used at 150 mg daily in adults >50 kg. While gastrointestinal and cutaneous side effects commonly occur at doses of 150 mg, adverse events occur less often at lower doses. We first reported erlotinib as effective for Olmsted syndrome, a rare hereditary EDD with painful PPK that results from variants in TRPV3. Erlotinib is now the treatment of choice for children and adults with Olmsted syndrome. Erlotinib is thought to inhibit formation of a complex that includes TRPV3, EGFR, and its primary skin-based ligand, TGF-a, which in turn regulates keratinocyte proliferation and differentiation. High-throughput screening to identify compounds that stabilize keratin filaments have also pointed to the EGFR pathway for targeting. Reviews and recent case reports have suggested the benefit of erlotinib for PC,

Given these preliminary data, we hypothesize that EGFR activation is a characteristic feature of keratinopathies. Further, we expect that oral low-dose erlotinib will improve the scaling and skin thickening of the spectrum of keratinopathies and be tolerated by most patients. For those who experience pain, particularly from plantar involvement, we predict that erlotinib therapy will improve mobility and pain. Finally, we aim to find the mechanism by which erlotinib improves the phenotypes of the various keratinopathies to better understand these disorders and predict response. We will look specifically at the impact on differentiation vs. hyperproliferation and barrier function, as well as the immune modulatory effects of the erlotinib using a multi-omics approach.

DETAILED DESCRIPTION:
We will conduct the first interventional multi-site Phase 1/2a trial of low-dose erlotinib to test its safety and efficacy as systemic treatment of moderate-to-severe keratinopathies.

The trial will have three parts:

During Part A, the natural history of keratinopathies and baseline for scores will be determined through at least 8 weeks of observation. We will use the mean of scores for our baseline, rather than a static measure at baseline to account for potential variability without the intervention.

Part B will be the dose escalation component, in which the subject will initiate 50 mg erlotinib,8 wks later escalate to 75 mg, and then 8 wks later to 100 mg erlotinib pending tolerance after each 8-week period. During this 24-week period, we will be assessing safety (Phase 1) in comparison to the 8-week baseline observation period (own control) and at ease dosing level. We will also evaluate efficacy based on dosing (Phase 2a) to achieve preliminary data to guide future trials if the use of erlotinib is a "go" based on safety.

Part C is the open-label extension period. Each participant will decide on the continued dosing for the subsequent 6 months in shared decision making with the investigator based on tolerance and effect. In total, the study involves 1 year on the erlotinib treatment, although the primary endpoint is 6 months after initiation. The additional 6 months will allow for further observation for potential toxicity and possible improved effect after additional time on drug. Participants will be eligible to participate in the open-label treatment period only if they have maintained >70% compliance with completion of studies during the initial 6 months.

ELIGIBILITY:
Inclusion Criteria:

The participant must be at least 18 years of age.

The participant must have a clinically and genetically confirmed diagnosis of a keratinopathy (Epidermolytic ichthyosis/EI: KRT 1, 2, or 10 pathogenic variant; Epidermolytic palmoplantar keratoderma/PPK: KRT 9; Pachyonychia congenita/PC form of PPK: KRT 6a, 6b, 6c, 16, 17). A blood or saliva sample will be collected for genetic confirmation if the underlying genetic change has not been confirmed by a CLIA-approved laboratory.

The participant must have an investigator scored IGA at screening and baseline of at least 2 (moderate) at affected sites.

The participant must abstain from use of any investigational drug or biologic within 4 weeks or 5 half-lives if longer, oral retinoid or oral steroid for at least 4 weeks, and topical medications (prescription or over-the-counter) in the week before the 8-week observation period. Otherwise stable medications (at least a month before the observation period and continued) will be allowed.

The participant agrees to use standard of care with respect to bathing and exfoliation/foot care, except in the week before the visits. Moisturizers/ emollients are allowed throughout the treatment period, but use must be consistent and withheld to the designated area of sampling on the arms (EI) or plantar foot (PC/PPK) for 48 hours prior to visits when skin samples are taken.

The participant is willing to have blood collected for safety and biopsies for investigation of mechanism.

Participant is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of the EI or PC/PPK.

Participant is able and willing to follow all study instructions

Exclusion Criteria:

The participant has EI or PC/PPK lesions on the assessment area that are infected or require therapy to treat the infection within 7 days of enrollment.

The participant has had major surgery during the past 4 weeks.

Participants have received an investigational drug or biologic within 4 weeks or 5 half-lives, whichever is longer, prior to starting treatment with and during treatment with erlotinib.

Participants must be off oral retinoid or oral steroid for at least 4 weeks before drug initiation.

Participants who require medications and OTC supplements that inhibit/ induce CYP3A4 activity to control concurrent medical conditions.

Participants with known hypersensitivity to any of the ingredients in the study medication formulation.

Participants previously treated for invasive cancer within the past 5 years unless the Investigator concludes history of cancer is not confounding to safety.

Participants who are pregnant, breastfeeding or planning to become pregnant during the study or within a month after the study ends.

Participants of childbearing potential who are unwilling or unable to comply with contraception measures.

The participant has any condition or situation which, in the Investigator's opinion, may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study.

Participants deemed by the investigator as unwilling or unable to remain compliant with all tests and procedures, adherence to the study drug administration regimen and other protocol-required activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Investigator Global Assessment (IGA) | 24 weeks
  Reduction in IGA score from baseline to week 24 of at least 50%. The Investigator Global Assessment/IGA will be the primary efficacy analysis, using the strata of clear 0, mild 1, moderate 2, severe 3, and very severe 4.
Percentage of Grade 3 and 4 Adverse Events | 24 weeks
  The percentage of participants with Grade 3 and 4 events, based on the current Common Toxicity Criteria for Adverse Events (CTCAE) listing

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, Principal Investigator — Northwestern University
Locations (1):
- Department of Dermatology, Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided